CLINICAL TRIAL: NCT04768608
Title: Clinical Trial for the Safety and Efficacy of Non-viral PD1 Integrated Anti-PSMA Chimeric Antigen Receptor T Cells in the Treatment of Refractory Castrate-Resistant Prostate Cancer
Brief Title: PD1 Integrated Anti-PSMA CART in Treating Patients With Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Bioray Laboratories (Industry)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-CAR-00CH2
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Castrate-Resistant Prostate Cancer
Keywords: Castrate-Resistant Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Group A: 0.5×10^6 cells / kg; Group B: 1.0×10^6 cells / kg; Group C: 2.0×10^6 cells / kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1-PSMA-CART (Experimental): Patients undergo leukapheresis by receiving cyclophosphamide and fludarabine on days -6 to -4, and then receive PD1-PSMA-CART intravenous injection (IV) at split doses from day 0 on.
  Interventions: Drug: PD1-PSMA-CART cells

INTERVENTIONS:
Drug: PD1-PSMA-CART cells — PD1-PSMA-CART cells will be given IV at split doses
  Other Names: Non-viral PD1 integrated anti-PSMA chimeric antigen receptor T cell

SUMMARY:
PD1-PSMA-CART in Treating Patients With Castrate-Resistant Prostate Cancer

DETAILED DESCRIPTION:
Clinical trial for the safety and efficacy of Non-viral programmed cell death protein-1(PD1) integrated anti-prostate-specific-membrane-antigen(PSMA) chimeric antigen receptor T(CART) cells in the treatment of Refractory Castrate-Resistant Prostate Cancer(CRPC)

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntarily sign informed consent.
* Aged 18 to 75 years old.
* Expected survival > 6 months.
* CRPC patients:Serum testosterone reached castration level (<50ng/dl or<1.7nmol/L) and: prostate specific antigen (PSA) increased more than 50% at intervals of one week or three consecutive times, with PSA>2 ng/ml; or imaging scans revealed two or more new lesions or enlargement of soft tissue lesions that met the criteria for evaluating solid tumor response.
* CRPC patients received abiraterone or chemotherapy for 3 months or more, and were ineffective or progressive (PSA continued to rise for 3 months, or bone scan/whole-body imaging showed local recurrence or new metastasis).
* Immunohistochemical staining of repetitive biopsy tissues showed the expression of PSMA in tumor cells was more than 50%.
* Eastern Cooperative Oncology Group (ECOG) score ≤2.
* Virological examination was negative.
* Hematological indexes: hemoglobin > 100 g/L, platelet count > 100×10^9/L, absolute neutrophil count > 1.5×10^9/L.

Exclusion Criteria:

* Prior treatment with any CART therapy targeting any target.
* Prior treatment with any PSMA targeting therapy.
* Need steroid therapy, except physiological replacement therapy.
* Prior treatment with any immunotherapy, including tumor vaccine therapy, radium-223, checkpoint inhibitors and others.
* Subjects with severe mental disorders.
* Subjects with other malignant tumors.
* Subjects with severe cardiovascular diseases: a, New York Heart Association (NYHA) stage III or IV congestive heart failure; b, history of myocardial infarction or coronary artery bypass grafting (CABG) within 6 months; c, clinical significance of ventricular arrhythmia, or history of unexplained syncope, non-vasovagal or dehydration; d, history of severe non-ischemic cardiomyopathy; e, the left ventricular ejection fraction (left ventricular ejection fraction< 55%) was decreased by echocardiography or multiple gated acquisition scan (within 8 weeks before peripheral blood mononuclear cell (PBMC) collection), and abnormal interventricular septal thickness and atrioventricular size associated with myocardial amyloidosis.
* Patients with ongoing or active infection.
* Organ function: a, Alanine aminotransferase or Aspartate aminotransferase >2.5*Upper limit of normal (ULN); Creatine kinase>1.5*ULN; Creatine kinase isoenzyme >1.5*ULN; Troponin T >1.5*ULN; b, Total bilirubin >1.5*ULN; c, Partial prothrombin time or activated partial thromboplastin time or international standardized ratio > 1.5*ULN without anticoagulant treatment.
* History of participation in other clinical studies within 3 months or treatment with any gene therapy product.
* Intolerant or allergic to cyclophosphamide or fludarabine.
* Subjects not appropriate to participate in this clinical study judged by investigators.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events | 28 days
  All adverse events (AEs) will be listed and summarized. Summaries of laboratory data will include, at a minimum, treatment-emergent laboratory abnormalities. Summaries of AEs and laboratory abnormalities will be based on the All Treated analysis set.

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) response rate | 180 days
  proportion of patients with ≥50% PSA decline from baseline at any time point after therapy and maintained for ≥4weeks
Radiographic response rate by RECIST 1.1 & PCWG3 | 180 days
  Proportion of patients with a best response of either complete response or partial response, assessed using Prostate Cancer Working group3(PCWG3) response criteria & Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Number of persistent CART cells detected by Quantitative Real-time Polymerase Chain Reaction or flow cytometry | 180 days
  Number of persistent CART cells detected by Quantitative Real-time Polymerase Chain Reaction or flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China